CLINICAL TRIAL: NCT00733902
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE
Brief Title: Tanezumab in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091011; P3 OA KNEE (Other: Alias Study Number)
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Arthritis; Osteoarthritis
Keywords: monoclonal antibody; RN624; PF-04383119; nerve growth factor; anti-nerve growth factor; OA; pain
MeSH Terms: conditions — Arthritis; Osteoarthritis; Hereditary Sensory and Autonomic Neuropathies; Pain | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tanezumab 10 mg (Experimental)
  Interventions: Biological: tanezumab
- Tanezumab 5 mg (Experimental)
  Interventions: Biological: tanezumab
- Tanezumab 2.5 mg (Experimental)
  Interventions: Biological: tanezumab
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: tanezumab — IV tanezumab 10 mg at 1 dose every 8 weeks
  Arms: Tanezumab 10 mg
Biological: tanezumab — IV tanezumab 5 mg at 1 dose every 8 weeks
  Arms: Tanezumab 5 mg
Biological: tanezumab — IV tanezumab 2.5 mg at 1 dose every 8 weeks
  Arms: Tanezumab 2.5 mg
Biological: Placebo — IV placebo to match tanezumab at 1 dose every 8 weeks
  Arms: Placebo

SUMMARY:
Test the efficacy and safety of 3 doses in Osteoarthritis of the knee in patients.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee according to ACR criteria with a Kellgren-Lawrence x-ray grade of 2.
* Unwilling or unable to take non-opiate pain medications, for whom non-opiate pain medications have not provided adequate pain relief or are candidates for knee injections arthroplasty or replace surgery.
* Pain level and function levels as required by the protocol at Screening and Baseline.
* Willing to discontinue pain medications (acetaminophen will be permitted up to a certain level) before and during the study.
* Must agree to the contraceptive requirements of the protocol if applicable.
* Must agree to the treatment plan, scheduled visits, and procedures of the protocol.

Exclusion Criteria:

* Pregnancy or intent to become pregnant during the study
* BMI greater than 39
* other severe pain, significant cardiac, neurological or psychological conditions, or above the protocol limits for laboratory and blood pressure results

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 697 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2009-08-24 (Actual); Study Completion 2010-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (82):
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Avail Clinical Rearch, LLC, DeLand, Florida
  - Avail Clinical Research, DeLand, Florida
  - Arthritis Associates of South Florida, Clinical Research Center, Delray Beach, Florida
  - Delray Research Associates, Delray Beach, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Neurorehabilitation & Diagnostic Services, Miami, Florida
  - Pharmax Research Clinic, LLC, Miami, Florida
  - South Medical Research Group, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - University Clinical Research Incorporated, Pembroke Pines, Florida
  - Advent Clinical Research Centers, Pinellas Park, Florida
  - AVIVOCLIN Clinical Services, Port Orange, Florida
  - Dale G. Bramlet, MD, P.L, St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Laureate Clinical Reseach Group, Atlanta, Georgia
  - Jefrey D. Lieberman, MD, PC, Decatur, Georgia
  - Early Family Practice Center, Fort Valley, Georgia
  - North Georgia Clinical Research, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - Sonora Clinical Research, Boise, Idaho
  - The Arthritis Center, Springfield, Illinois
  - Memorial Health System, Inc./ Michiana Arthritis & Osteoporosis Center, South Bend, Indiana
  - Memorial Health System, Inc., South Bend, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Arthritis Center of Lexington, Lexington, Kentucky
  - Bluegrass Community Research, Inc, Lexington, Kentucky
  - David H. Neustadt P.S.C., Louisville, Kentucky
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - The Baton Rouge Clinic, Baton Rouge, Louisiana
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Office of Peter A. Holt, MD, Baltimore, Maryland
  - The Arthritis and Osteoporosis Center of Maryland, Frederick, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Mansfield Health Center, Mansfield, Massachusetts
  - Arthritis Associates Inc., Peabody, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Ann Arbor Clinical Research, Ann Arbor, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - MAPS Applied Research Center, Edina, Minnesota
  - Medical Advanced Pain Specialists, Edina, Minnesota
  - Mercy Health Research, St Louis, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Incorporated, Albuquerque, New Mexico
  - Health Sciences Research Center at Asthma & Allergy Assoc., PC, Elmira, New York
  - Health Sciences Research Center at Asthma and Allergy Associates P.C., Ithaca, New York
  - The Medical Research Network, LLC, New York, New York
  - Prem C. Chatpar, MD, LLC, Plainview, New York
  - AAIR Research Center, Rochester, New York
  - Arthristis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - C.A.R.E. Center, Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Hilltop Physicians Inc, Hightop Medical Research Center, Cincinnati, Ohio
  - Southwest Rheumatology and Research Group, LLC, Middleburg Heights, Ohio
  - Pharmacotherapy Research Associates,Inc, Zanesville, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - EPIC Imaging West, Beaverton, Oregon
  - EPIC Imaging East:, Portland, Oregon
  - Covance CRU, Inc., Portland, Oregon
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Appalachian Medical Research, Johnson City, Tennessee
  - Walter Chase, MD, Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Radiant Research, San Antonio, Texas
  - Texas Arthritis Research Center, PA, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Clinical Trials Northwest, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Hochberg MC, Tive LA, Abramson SB, Vignon E, Verburg KM, West CR, Smith MD, Hungerford DS. When Is Osteonecrosis Not Osteonecrosis?: Adjudication of Reported Serious Adverse Joint Events in the Tanezumab Clinical Development Program. Arthritis Rheumatol. 2016 Feb;68(2):382-91. doi: 10.1002/art.39492. PMID 26554876
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091011&StudyName=Tanezumab%20in%20Osteoarthritis%20of%20the%20Knee%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who discontinued due to lack of efficacy or completed the treatment in this study were eligible to enroll in safety extension study A4091016 (NCT00809783).
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 milligram (mg) intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Started | 174 | 174 | 174 | 175
Treated | 172 | 172 | 172 | 174
Completed | 10 | 12 | 13 | 11
Not Completed | 164 | 162 | 161 | 164
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Adverse Event | 3 | 4 | 7 | 11
Not completed — Lack of Efficacy | 56 | 21 | 34 | 23
Not completed — Protocol Violation | 4 | 6 | 3 | 3
Not completed — Withdrawal by Subject | 10 | 5 | 4 | 16
Not completed — Entered extension study | 89 | 124 | 111 | 109
Not completed — Randomized but not treated | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg | Total
Number analyzed (Participants) | 172 | 172 | 172 | 174 | 690
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.9) | 60.8 (9.8) | 62.1 (10.5) | 61.4 (10.5) | 61.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 94 | 101 | 106 | 420
  Male | 53 | 78 | 71 | 68 | 270

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA). WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain.
Time Frame: Baseline (Day 1), Week 16
Population: Modified intent-to-treat (mITT) analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded and from site 1006. BOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline | 7.05 (1.45) | 7.16 (1.44) | 7.19 (1.41) | 6.99 (1.43)
  Change at Week 16 | -2.51 (2.63) | -3.27 (2.78) | -3.39 (2.65) | -3.67 (2.83)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Analysis of Covariance (ANCOVA) was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.015, ANCOVA; Least Squares (LS) Mean Difference = -0.73, 95% CI 2-sided [-1.32 to -0.14], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-1.43 to -0.25], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.20, 95% CI 2-sided [-1.78 to -0.61], Standard Error of Mean 0.30

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC physical function is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index knee during past 48 hours. It is calculated as mean of the scores from 17 individual questions, each scored on a NRS of 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicate worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 16
Population: mITT analysis set. BOCF method was used to impute missing values. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 155 | 154
units on a scale
  Baseline | 6.64 (1.59) | 6.86 (1.58) | 6.91 (1.49) | 6.69 (1.62)
  Change at Week 16 | -2.06 (2.45) | -2.93 (2.67) | -3.14 (2.59) | -3.34 (2.70)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.009, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.32 to -0.19], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.54 to -0.41], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.24, 95% CI 2-sided [-1.80 to -0.68], Standard Error of Mean 0.28

3. Primary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 16: Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all the ways your osteoarthritis in your knee affects you, how are you doing today?". Participants responded on a scale ranging from 1-5, where 1= very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5= very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Week 16
Population: mITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded and from site 1006. BOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline | 3.40 (0.58) | 3.47 (0.63) | 3.45 (0.63) | 3.45 (0.59)
  Change at Week 16 | -0.51 (0.83) | -0.87 (0.93) | -0.91 (0.95) | -1.05 (1.06)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.52 to -0.13], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.56 to -0.17], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-0.70 to -0.31], Standard Error of Mean 0.10

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 2, 4, 8, 12, 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Change at Week 2 | -2.75 (2.46) | -3.08 (2.55) | -2.52 (2.39) | -2.68 (2.56)
  Change at Week 4 | -2.72 (2.39) | -3.70 (2.63) | -3.44 (2.40) | -3.72 (2.58)
  Change at Week 8 | -2.53 (2.46) | -3.40 (2.54) | -3.32 (2.38) | -3.84 (2.56)
  Change at Week 12 | -2.55 (2.59) | -3.70 (2.70) | -3.51 (2.70) | -3.80 (2.69)
  Change at Week 24 | -2.39 (2.63) | -3.10 (2.84) | -2.99 (2.64) | -3.55 (2.91)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 2: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.326, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.80 to 0.27], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.275, ANCOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-0.24 to 0.83], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.918, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.51 to 0.56], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 4: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.93, 95% CI 2-sided [-1.47 to -0.40], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.013, ANCOVA; LS Mean Difference = -0.68, 95% CI 2-sided [-1.22 to -0.15], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.03, 95% CI 2-sided [-1.57 to -0.49], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 8: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.82, 95% CI 2-sided [-1.36 to -0.28], Standard Error of Mean 0.27
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.006, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.29 to -0.21], Standard Error of Mean 0.27
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.33, 95% CI 2-sided [-1.87 to -0.79], Standard Error of Mean 0.27
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 12: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.10, 95% CI 2-sided [-1.68 to -0.53], Standard Error of Mean 0.29
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.91, 95% CI 2-sided [-1.48 to -0.33], Standard Error of Mean 0.29
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.29, 95% CI 2-sided [-1.87 to -0.72], Standard Error of Mean 0.29
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 24: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.027, ANCOVA; LS Mean Difference = -0.68, 95% CI 2-sided [-1.28 to -0.08], Standard Error of Mean 0.31
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.071, ANCOVA; LS Mean Difference = -0.55, 95% CI 2-sided [-1.15 to 0.05], Standard Error of Mean 0.31
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.18, 95% CI 2-sided [-1.78 to -0.58], Standard Error of Mean 0.31

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 2, 4, 8, 12, 16, 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 4
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded and from site 1006. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline | 7.05 (1.45) | 7.16 (1.44) | 7.19 (1.41) | 6.99 (1.43)
  Change at Week 2 | -2.75 (2.46) | -3.08 (2.55) | -2.52 (2.39) | -2.68 (2.56)
  Change at Week 4 | -2.89 (2.44) | -3.81 (2.57) | -3.45 (2.40) | -3.82 (2.54)
  Change at Week 8 | -2.65 (2.44) | -3.44 (2.53) | -3.44 (2.32) | -4.01 (2.47)
  Change at Week 12 | -2.95 (2.51) | -3.96 (2.53) | -3.77 (2.56) | -4.13 (2.49)
  Change at Week 16 | -2.89 (2.57) | -3.46 (2.69) | -3.60 (2.54) | -4.17 (2.55)
  Change at Week 24 | -2.93 (2.59) | -3.38 (2.72) | -3.40 (2.57) | -4.11 (2.67)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.326, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.80 to 0.27], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.275, ANCOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-0.24 to 0.83], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.918, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.51 to 0.56], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.85, 95% CI 2-sided [-1.39 to -0.32], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.052, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-1.06 to 0.00], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.50 to -0.44], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.006, ANCOVA; LS Mean Difference = -0.74, 95% CI 2-sided [-1.26 to -0.21], Standard Error of Mean 0.27
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -0.76, 95% CI 2-sided [-1.28 to -0.24], Standard Error of Mean 0.27
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.38, 95% CI 2-sided [-1.91 to -0.86], Standard Error of Mean 0.27
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.96, 95% CI 2-sided [-1.50 to -0.43], Standard Error of Mean 0.27
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -0.77, 95% CI 2-sided [-1.30 to -0.23], Standard Error of Mean 0.27
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.22, 95% CI 2-sided [-1.75 to -0.69], Standard Error of Mean 0.27
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 16: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.061, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-1.07 to 0.02], Standard Error of Mean 0.28
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.021, ANCOVA; LS Mean Difference = -0.65, 95% CI 2-sided [-1.20 to -0.10], Standard Error of Mean 0.28
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.30, 95% CI 2-sided [-1.85 to -0.76], Standard Error of Mean 0.28
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.166, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.95 to 0.16], Standard Error of Mean 0.28
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.167, ANOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.95 to 0.16], Standard Error of Mean 0.28
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.20, 95% CI 2-sided [-1.75 to -0.64], Standard Error of Mean 0.28

6. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 2, 4, 8, 12, 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC physical function is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint during past 48 hours. It is calculated as mean of the scores from 17 individual questions, each scored on a NRS of 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicate worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living
Time Frame: Baseline, Week 2, 4, 8, 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 155 | 154
units on a scale
  Change at Week 2 | -2.17 (2.40) | -2.85 (2.62) | -2.34 (2.27) | -2.61 (2.57)
  Change at Week 4 | -2.13 (2.36) | -3.23 (2.66) | -3.09 (2.35) | -3.41 (2.56)
  Change at Week 8 | -2.00 (2.31) | -2.97 (2.58) | -2.98 (2.36) | -3.47 (2.58)
  Change at Week 12 | -2.13 (2.50) | -3.38 (2.64) | -3.25 (2.62) | -3.51 (2.66)
  Change at Week 24 | -2.01 (2.44) | -2.77 (2.71) | -2.74 (2.61) | -3.23 (2.83)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.044, ANCOVA; LS Mean Difference = -0.54, 95% CI 2-sided [-1.07 to -0.02], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.875, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.57 to 0.48], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.129, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.93 to 0.12], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.51 to -0.45], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.85, 95% CI 2-sided [-1.38 to -0.32], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.23, 95% CI 2-sided [-1.76 to -0.70], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.83, 95% CI 2-sided [-1.35 to -0.30], Standard Error of Mean 0.27
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.87, 95% CI 2-sided [-1.39 to -0.34], Standard Error of Mean 0.27
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.42, 95% CI 2-sided [-1.94 to -0.90], Standard Error of Mean 0.27
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.14, 95% CI 2-sided [-1.70 to -0.58], Standard Error of Mean 0.29
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.01, 95% CI 2-sided [-1.57 to -0.45], Standard Error of Mean 0.29
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.35, 95% CI 2-sided [-1.91 to -0.79], Standard Error of Mean 0.28
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.021, ANCOVA; LS Mean Difference = -0.68, 95% CI 2-sided [-1.26 to -0.10], Standard Error of Mean 0.29
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.029, ANCOVA; LS Mean Difference = -0.64, 95% CI 2-sided [-1.22 to -0.07], Standard Error of Mean 0.29
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.20, 95% CI 2-sided [-1.78 to -0.62], Standard Error of Mean 0.29

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 2, 4, 8, 12, 16, 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 6
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set. LOCF method was used to impute missing values. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 155 | 154
units on a scale
  Baseline | 6.64 (1.59) | 6.86 (1.58) | 6.91 (1.49) | 6.69 (1.62)
  Change at Week 2 | -2.17 (2.40) | -2.85 (2.62) | -2.34 (2.27) | -2.61 (2.57)
  Change at Week 4 | -2.27 (2.46) | -3.36 (2.59) | -3.16 (2.32) | -3.51 (2.54)
  Change at Week 8 | -2.06 (2.36) | -3.01 (2.55) | -3.12 (2.31) | -3.64 (2.51)
  Change at Week 12 | -2.39 (2.52) | -3.55 (2.53) | -3.49 (2.52) | -3.80 (2.49)
  Change at Week 16 | -2.33 (2.47) | -3.04 (2.60) | -3.31 (2.53) | -3.81 (2.47)
  Change at Week 24 | -2.35 (2.55) | -2.96 (2.63) | -3.11 (2.62) | -3.78 (2.62)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.044, ANCOVA; LS Mean Difference = -0.54, 95% CI 2-sided [-1.07 to -0.02], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.875, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.57 to 0.48], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.129, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.93 to 0.12], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.94, 95% CI 2-sided [-1.46 to -0.41], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.004, ANCOVA; L Mean Difference = -0.76, 95% CI 2-sided [-1.28 to -0.24], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.19, 95% CI 2-sided [-1.71 to -0.67], Standard Error of Mean 0.26
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.82, 95% CI 2-sided [-1.33 to -0.30], Standard Error of Mean 0.26
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.95, 95% CI 2-sided [-1.46 to -0.43], Standard Error of Mean 0.26
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.53, 95% CI 2-sided [-2.04 to -1.02], Standard Error of Mean 0.26
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.03, 95% CI 2-sided [-1.56 to -0.51], Standard Error of Mean 0.27
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.99, 95% CI 2-sided [-1.52 to -0.46], Standard Error of Mean 0.27
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.37, 95% CI 2-sided [-1.90 to -0.85], Standard Error of Mean 0.27
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.030, ANCOVA; LS Mean Difference = -0.59, 95% CI 2-sided [-1.12 to -0.06], Standard Error of Mean 0.27
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.86, 95% CI 2-sided [-1.39 to -0.32], Standard Error of Mean 0.27
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.43, 95% CI 2-sided [-1.96 to -0.90], Standard Error of Mean 0.27
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.085, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-1.03 to 0.07], Standard Error of Mean 0.28
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.026, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-1.18 to -0.08], Standard Error of Mean 0.28
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.39, 95% CI 2-sided [-1.94 to -0.84], Standard Error of Mean 0.28

8. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscales at Week 2, 4, 8, 12, 16, 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in index knee during past 48 hours. It is calculated as mean of the scores from 2 individual questions scored on NRS of (no stiffness) to 10 (extreme stiffness), with higher scores indicate higher stiffness. Total score range for WOMAC stiffness subscale score is (no stiffness) to 10 (extreme stiffness), where higher scores indicate higher stiffness. Stiffness is defined as a sensation of decreased ease in movement of knee.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline | 6.94 (1.80) | 6.98 (1.90) | 7.05 (1.69) | 6.89 (2.04)
  Change at Week 2 | -2.09 (2.53) | -2.91 (2.79) | -2.50 (2.60) | -2.70 (2.82)
  Change at Week 4 | -2.12 (2.46) | -3.33 (2.79) | -3.28 (2.62) | -3.54 (2.75)
  Change at Week 8 | -1.98 (2.48) | -2.91 (2.83) | -3.06 (2.55) | -3.70 (2.75)
  Change at Week 12 | -2.10 (2.60) | -3.44 (2.94) | -3.38 (2.82) | -3.75 (2.92)
  Change at Week 16 | -2.06 (2.47) | -2.95 (2.92) | -3.20 (2.72) | -3.50 (2.92)
  Change at Week 24 | -2.02 (2.49) | -2.86 (2.87) | -2.68 (2.70) | -3.44 (3.03)

9. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 2, 4, 8, 12, 16, 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 8
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline | 6.94 (1.80) | 6.98 (1.90) | 7.05 (1.69) | 6.89 (2.04)
  Change at Week 2 | -2.09 (2.53) | -2.91 (2.79) | -2.50 (2.60) | -2.70 (2.82)
  Change at Week 4 | -2.31 (2.52) | -3.44 (2.71) | -3.32 (2.61) | -3.66 (2.79)
  Change at Week 8 | -2.11 (2.47) | -2.96 (2.80) | -3.22 (2.47) | -3.83 (2.72)
  Change at Week 12 | -2.42 (2.57) | -3.59 (2.82) | -3.62 (2.72) | -4.04 (2.79)
  Change at Week 16 | -2.40 (2.45) | -3.07 (2.86) | -3.36 (2.67) | -3.99 (2.75)
  Change at Week 24 | -2.45 (2.55) | -3.07 (2.77) | -3.07 (2.71) | -3.94 (2.88)

10. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 2, 4, 8, 12, 24: Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all the ways your osteoarthritis in your knee affects you, how are you doing today". Participants responded on a scale ranging from 1-5, where 1= very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5= very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Week 2, 4, 8, 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Change at Week 2 | -0.55 (0.87) | -0.91 (0.90) | -0.63 (0.88) | -0.82 (0.99)
  Change at Week 4 | -0.55 (0.78) | -1.04 (0.92) | -1.04 (0.91) | -1.16 (0.99)
  Change at Week 8 | -0.46 (0.73) | -0.84 (0.90) | -0.84 (0.91) | -1.16 (0.99)
  Change at Week 12 | -0.53 (0.82) | -1.01 (0.98) | -0.94 (0.89) | -1.17 (1.03)
  Change at Week 24 | -0.53 (0.83) | -0.77 (0.90) | -0.70 (0.94) | -0.93 (1.11)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.49 to -0.14], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.486, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.24 to 0.11], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.42 to -0.06], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.63 to -0.26], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.64 to -0.28], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.76 to -0.39], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.53 to -0.16], Standard Error of Mean 0.09
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.54 to -0.17], Standard Error of Mean 0.09
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.67, 95% CI 2-sided [-0.85 to -0.49], Standard Error of Mean 0.09
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.63 to -0.25], Standard Error of Mean 0.10
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.57 to -0.19], Standard Error of Mean 0.10
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.61, 95% CI 2-sided [-0.80 to -0.42], Standard Error of Mean 0.10
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.035, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.42 to -0.02], Standard Error of Mean 0.10
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.125, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.36 to 0.04], Standard Error of Mean 0.10
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.58 to -0.18], Standard Error of Mean 0.10

11. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 2, 4, 8, 12, 16, 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 10
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline | 3.40 (0.58) | 3.47 (0.63) | 3.45 (0.63) | 3.45 (0.59)
  Change at Week 2 | -0.55 (0.87) | -0.91 (0.90) | -0.63 (0.88) | -0.82 (0.99)
  Change at Week 4 | -0.57 (0.83) | -1.08 (0.91) | -1.05 (0.91) | -1.18 (1.00)
  Change at Week 8 | -0.47 (0.79) | -0.86 (0.90) | -0.90 (0.92) | -1.21 (0.98)
  Change at Week 12 | -0.60 (0.88) | -1.05 (0.97) | -0.99 (0.90) | -1.28 (1.03)
  Change at Week 16 | -0.58 (0.91) | -0.90 (0.93) | -0.97 (0.96) | -1.19 (1.05)
  Change at Week 24 | -0.60 (0.92) | -0.82 (0.90) | -0.82 (1.00) | -1.13 (1.12)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.49 to -0.14], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.486, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.24 to 0.11], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.42 to -0.06], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.64 to -0.28], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.62 to -0.26], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.75 to -0.39], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.53 to -0.16], Standard Error of Mean 0.09
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.58 to -0.22], Standard Error of Mean 0.09
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.71, 95% CI 2-sided [-0.89 to -0.52], Standard Error of Mean 0.09
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.59 to -0.22], Standard Error of Mean 0.09
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.55 to -0.18], Standard Error of Mean 0.09
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.65, 95% CI 2-sided [-0.83 to -0.46], Standard Error of Mean 0.09
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.47 to -0.09], Standard Error of Mean 0.10
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.55 to -0.17], Standard Error of Mean 0.10
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-0.77 to -0.39], Standard Error of Mean 0.10
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.090, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.37 to 0.03], Standard Error of Mean 0.10
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.053, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.39 to 0.00], Standard Error of Mean 0.10
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.50, 95% CI 2-sided [-0.70 to -0.30], Standard Error of Mean 0.10

12. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Response: Baseline Observation Carried Forward (BOCF)
Description: OMERACT-OARSI response: greater than or equal to (>=) 50 percent (%) improvement from baseline and absolute change from baseline of >=2 units at Week of interest in WOMAC pain or physical function subscale, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit at Week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Week 2 | 62.3 | 68.2 | 60.9 | 68.2
  Week 4 | 57.1 | 70.8 | 75.0 | 77.3
  Week 8 | 52.6 | 72.1 | 73.7 | 78.6
  Week 12 | 53.2 | 74.7 | 74.4 | 77.9
  Week 16 | 53.9 | 68.2 | 69.9 | 70.8
  Week 24 | 51.3 | 62.3 | 64.1 | 69.5

13. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Response: Last Observation Carried Forward (LOCF)
Description: OMERACT-OARSI response: >= 50% improvement from baseline and absolute change from baseline of >=2 units at Week of interest in WOMAC pain or physical function subscale, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit at Week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Week 2 | 62.3 | 68.2 | 60.9 | 68.2
  Week 4 | 61.7 | 74.0 | 76.3 | 80.5
  Week 8 | 57.1 | 73.4 | 77.6 | 83.1
  Week 12 | 64.9 | 80.5 | 81.4 | 85.7
  Week 16 | 65.6 | 72.7 | 75.6 | 82.5
  Week 24 | 65.6 | 70.8 | 75.0 | 82.5

14. Secondary Outcome: Percentage of Participants With at Least 30% and 50% Reduction From Baseline in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 4
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Week 2: >=30% reduction | 57.8 | 60.4 | 50.6 | 55.2
  Week 2: >=50% reduction | 40.9 | 44.8 | 32.1 | 41.6
  Week 4: >=30% reduction | 57.1 | 66.2 | 66.7 | 72.1
  Week 4: >=50% reduction | 40.3 | 56.5 | 50.6 | 57.8
  Week 8: >=30% reduction | 50.0 | 65.6 | 67.9 | 74.0
  Week 8: >=50% reduction | 38.3 | 48.7 | 50.0 | 63.6
  Week 12: >=30% reduction | 52.6 | 67.5 | 66.0 | 73.4
  Week 12: >=50% reduction | 39.0 | 57.1 | 56.4 | 57.8
  Week 16: >=30% reduction | 51.3 | 64.3 | 65.4 | 68.2
  Week 16: >=50% reduction | 39.0 | 50.6 | 50.0 | 61.7
  Week 24: >=30% reduction | 48.7 | 59.7 | 59.6 | 66.9
  Week 24: >=50% reduction | 40.3 | 47.4 | 44.9 | 57.1

15. Secondary Outcome: Percentage of Participants With at Least 30 Percent (%) and 50% Reduction From Baseline in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score: Last Observation Carried Forward (LOCF)
Description: as for outcome 4
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Week 2: >=30% reduction | 57.8 | 60.4 | 50.6 | 55.2
  Week 2: >=50% reduction | 40.9 | 44.8 | 32.1 | 41.6
  Week 4: >=30% reduction | 60.4 | 69.5 | 67.3 | 74.7
  Week 4: >=50% reduction | 42.2 | 57.8 | 50.6 | 59.1
  Week 8: >=30% reduction | 53.9 | 66.9 | 71.2 | 77.9
  Week 8: >=50% reduction | 39.0 | 49.4 | 51.3 | 65.6
  Week 12: >=30% reduction | 63.0 | 73.4 | 72.4 | 79.9
  Week 12: >=50% reduction | 42.9 | 60.4 | 58.3 | 61.7
  Week 16: >=30% reduction | 61.7 | 68.8 | 70.5 | 78.6
  Week 16: >=50% reduction | 42.2 | 53.2 | 51.3 | 68.2
  Week 24: >=30% reduction | 61.0 | 66.2 | 68.6 | 78.6
  Week 24: >=50% reduction | 44.8 | 51.9 | 49.4 | 64.9

16. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement From Baseline in Patient Global Assessment (PGA) of Osteoarthritis: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 10
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Week 2 | 11.7 | 24.0 | 14.7 | 21.4
  Week 4 | 10.4 | 31.8 | 24.4 | 37.7
  Week 8 | 9.1 | 23.4 | 19.9 | 33.8
  Week 12 | 15.6 | 32.5 | 24.4 | 39.6
  Week 16 | 13.6 | 24.7 | 23.7 | 30.5
  Week 24 | 16.2 | 20.8 | 18.6 | 32.5

17. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement From Baseline in Patient Global Assessment (PGA) of Osteoarthritis: Last Observation Carried Forward (LOCF)
Description: as for outcome 10
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Week 2 | 11.7 | 24.0 | 14.7 | 21.4
  Week 4 | 11.7 | 32.5 | 24.4 | 38.3
  Week 8 | 10.4 | 23.4 | 21.2 | 35.7
  Week 12 | 17.5 | 33.1 | 25.0 | 42.9
  Week 16 | 15.6 | 25.3 | 25.0 | 35.7
  Week 24 | 18.8 | 21.4 | 21.8 | 39.6

18. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline to Week 16 in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Participants with specified reduction (as percent) from baseline up to Week 16 are reported.
Time Frame: Baseline up to Week 16
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Greater than (>) 0% | 61.0 | 79.2 | 79.5 | 76.0
  >=10% | 59.7 | 75.3 | 78.2 | 74.7
  >=20% | 54.5 | 70.8 | 69.9 | 70.1
  >=30% | 51.3 | 64.3 | 65.4 | 68.2
  >=40% | 48.7 | 58.4 | 57.7 | 67.5
  >=50% | 67.5 | 50.6 | 50.0 | 61.7
  >=60% | 31.8 | 39.0 | 45.5 | 55.8
  >=70% | 23.4 | 33.1 | 39.1 | 44.2
  >=80% | 13.6 | 27.3 | 27.6 | 31.8
  >=90% | 5.2 | 14.9 | 12.8 | 24.0
  =100% | 0.1 | 4.5 | 5.8 | 7.1

19. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline to Week 16 in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score: Last Observation Carried Forward (LOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee during past 48 hours. It is calculated as mean of the scores from 5 individual questions, each scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (extreme pain), where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. Participants with specified reduction (as percent) from baseline up to Week 16 are reported.
Time Frame: Baseline up to Week 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  >0% | 84.4 | 87.7 | 92.9 | 92.9
  >=10% | 77.9 | 83.1 | 87.2 | 90.9
  >=20% | 66.2 | 76.6 | 75.6 | 83.1
  >=30% | 61.7 | 68.8 | 70.5 | 78.6
  >=40% | 55.2 | 62.3 | 60.3 | 75.3
  >=50% | 42.2 | 53.2 | 51.3 | 68.2
  >=60% | 33.8 | 40.9 | 46.2 | 62.3
  >=70% | 24.7 | 33.8 | 39.7 | 47.4
  >=80% | 14.3 | 27.3 | 28.2 | 34.4
  >=90% | 5.8 | 14.9 | 13.5 | 25.3
  =100% | 0.1 | 4.5 | 5.8 | 8.4

20. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Knee at Week 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24: Baseline Observation Carried Forward (BOCF)
Description: Participants assessed daily average knee pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst pain). Baseline score was calculated as the mean of the scores over the 3 days and a weekly mean was calculated using the daily pain scores within each study week. The change from Baseline was calculated using difference between each post-baseline weekly mean and the Baseline mean score.
Time Frame: Baseline, Week 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 153 | 152 | 151 | 153
units on a scale
  Baseline | 6.38 (1.93) | 6.70 (1.83) | 6.74 (1.63) | 6.55 (1.91)
  Change at Week 1 | -1.21 (1.97) | -1.87 (2.04) | -1.83 (1.84) | -2.09 (2.03)
  Change at Week 2 | -1.68 (2.21) | -2.12 (2.42) | -1.83 (2.02) | -2.15 (2.31)
  Change at Week 3 | -1.73 (2.22) | -2.38 (2.52) | -1.90 (2.06) | -2.17 (2.47)
  Change at Week 4 | -1.81 (2.32) | -2.73 (2.49) | -2.47 (2.14) | -2.99 (2.52)
  Change at Week 6 | -1.83 (2.37) | -2.78 (2.66) | -2.50 (2.20) | -3.07 (2.59)
  Change at Week 8 | -1.67 (2.28) | -2.45 (2.61) | -2.47 (2.18) | -3.10 (2.63)
  Change at Week 10 | -1.84 (2.41) | -2.80 (2.76) | -2.65 (2.40) | -3.33 (2.82)
  Change at Week 12 | -1.82 (2.37) | -2.91 (2.76) | -2.78 (2.52) | -3.27 (2.72)
  Change at Week 16 | -1.73 (2.34) | -2.28 (2.69) | -2.58 (2.47) | -3.15 (2.76)
  Change at Week 20 | -1.80 (2.30) | -2.80 (2.88) | -2.81 (2.54) | -3.27 (2.83)
  Change at Week 24 | -1.63 (2.21) | -2.44 (2.78) | -2.29 (2.48) | -2.98 (2.93)

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 2, 4, 8, 12, 16, 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis of knee. WOMAC average score is the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, where higher score indicates worse response.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline | 6.88 (1.43) | 7.00 (1.46) | 7.05 (1.38) | 6.86 (1.52)
  Change at Week 2 | -2.34 (2.31) | -2.95 (2.53) | -2.46 (2.29) | -2.67 (2.49)
  Change at Week 4 | -2.32 (2.28) | -3.42 (2.58) | -3.29 (2.35) | -3.55 (2.50)
  Change at Week 8 | -2.17 (2.28) | -3.09 (2.53) | -3.13 (2.31) | -3.68 (2.52)
  Change at Week 12 | -2.26 (2.46) | -3.51 (2.65) | -3.38 (2.62) | -3.70 (2.64)
  Change at Week 16 | -2.21 (2.41) | -3.05 (2.67) | -3.25 (2.56) | -3.51 (2.71)
  Change at Week 24 | -2.14 (2.40) | -2.91 (2.70) | -2.81 (2.56) | -3.43 (2.82)

22. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item at Week 2, 4, 8, 12, 16, 24: Baseline Observation Carried Forward (BOCF)
Description: Participants answered, Question (Q)1: "How much pain have you had when walking on a flat surface?" and Q2: "How much pain have you had when going up or down the stairs?". Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set. BOCF method was used to impute missing values. Here, 'Number Analyzed' signifies participants evaluated at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline: Q1 | 6.90 (1.67) | 7.18 (1.72) | 7.28 (1.59) | 6.96 (1.71)
  Baseline: Q2: number analyzed (Participants) | 152 | 154 | 155 | 154
  Baseline: Q2 | 8.10 (1.45) | 8.21 (1.55) | 8.21 (1.45) | 8.18 (1.44)
  Change at Week 2: Q1 | -2.44 (2.58) | -3.23 (2.87) | -2.58 (2.56) | -2.95 (2.73)
  Change at Week 2: Q2: number analyzed (Participants) | 152 | 154 | 155 | 154
  Change at Week 2: Q2 | -2.49 (2.57) | -3.08 (2.84) | -2.59 (2.48) | -2.99 (2.66)
  Change at Week 4: Q1 | -2.55 (2.50) | -3.78 (2.90) | -3.49 (2.49) | -3.89 (2.66)
  Change at Week 4: Q2: number analyzed (Participants) | 152 | 154 | 155 | 154
  Change at Week 4: Q2 | -2.54 (2.53) | -3.67 (2.96) | -3.43 (2.60) | -3.94 (2.80)
  Change at Week 8: Q1 | -2.41 (2.64) | -3.40 (2.95) | -3.30 (2.45) | -3.86 (2.73)
  Change at Week 8: Q2: number analyzed (Participants) | 152 | 154 | 155 | 154
  Change at Week 8: Q2 | -2.34 (2.50) | -3.28 (2.91) | -3.26 (2.52) | -3.95 (2.87)
  Change at Week 12: Q1 | -2.38 (2.65) | -3.73 (2.98) | -3.51 (2.82) | -3.75 (2.80)
  Change at Week 12: Q2: number analyzed (Participants) | 152 | 154 | 155 | 154
  Change at Week 12: Q2 | -2.42 (2.67) | -3.77 (3.08) | -3.48 (3.00) | -3.95 (3.04)
  Change at Week 16: Q1 | -2.44 (2.73) | -3.26 (3.00) | -3.42 (2.84) | -3.64 (2.99)
  Change at Week 16: Q2: number analyzed (Participants) | 152 | 154 | 155 | 154
  Change at Week 16: Q2 | -2.28 (2.55) | -3.23 (3.00) | -3.37 (2.86) | -3.79 (3.02)
  Change at Week 24: Q1 | -2.27 (2.66) | -3.10 (3.08) | -3.03 (2.80) | -3.56 (3.13)
  Change at Week 24: Q2: number analyzed (Participants) | 152 | 154 | 155 | 154
  Change at Week 24: Q2 | -2.13 (2.68) | -3.10 (3.09) | -2.97 (2.89) | -3.75 (3.07)

23. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 12, 24: Baseline Observation Carried Forward (BOCF)
Description: SF-36v2: standardized survey evaluating 8 domains of functional health and wellbeing (physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health). Total score for each domain were scaled 0 (poor health) to 100 (best health), higher scores indicating good health condition.
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
units on a scale
  Baseline: General health | 67.16 (18.72) | 65.39 (17.74) | 65.99 (17.82) | 69.38 (17.47)
  Baseline: Physical Function | 32.64 (19.16) | 30.52 (20.07) | 30.46 (19.11) | 33.42 (20.90)
  Baseline: Role Physical | 45.74 (25.76) | 42.25 (24.41) | 43.51 (24.39) | 45.33 (27.98)
  Baseline: Bodily Pain | 34.48 (15.60) | 33.84 (17.50) | 33.50 (16.28) | 34.20 (16.06)
  Baseline: Vitality | 51.42 (19.22) | 54.26 (18.62) | 55.25 (18.27) | 53.45 (21.43)
  Baseline: Social Function | 69.48 (25.53) | 68.91 (27.28) | 70.03 (25.59) | 72.65 (24.58)
  Baseline: Role Emotional | 73.43 (27.13) | 67.48 (29.88) | 71.85 (28.29) | 71.37 (30.19)
  Baseline: Mental Health | 74.35 (16.18) | 75.49 (18.23) | 76.44 (16.86) | 76.36 (17.42)
  Change at Week 12: General health | 3.28 (12.12) | 3.62 (11.81) | 5.81 (14.17) | 5.11 (13.44)
  Change at Week 12: Physical Function | 8.26 (18.75) | 19.99 (22.43) | 18.12 (22.72) | 19.34 (22.36)
  Change at Week 12: Role Physical | 8.97 (24.21) | 19.85 (27.50) | 19.51 (25.54) | 18.06 (25.56)
  Change at Week 12: Bodily Pain | 11.83 (19.60) | 22.46 (25.53) | 21.19 (23.77) | 24.36 (24.62)
  Change at Week 12: Vitality | 4.34 (14.62) | 6.94 (16.16) | 6.69 (18.58) | 9.28 (17.04)
  Change at Week 12: Social Function | 6.25 (22.20) | 10.96 (25.70) | 11.46 (21.15) | 7.47 (22.44)
  Change at Week 12: Role Emotional | 5.30 (21.28) | 10.71 (26.47) | 8.81 (23.95) | 10.50 (28.26)
  Change at Week 12: Mental Health | 3.80 (13.59) | 3.41 (14.08) | 4.17 (15.91) | 3.77 (14.02)
  Change at Week 24: General health | 3.38 (11.81) | 4.27 (11.87) | 3.31 (13.10) | 2.94 (10.20)
  Change at Week 24: Physical Function | 8.75 (19.53) | 15.25 (20.98) | 13.54 (23.00) | 17.97 (23.32)
  Change at Week 24: Role Physical | 7.75 (22.97) | 14.12 (26.73) | 12.82 (23.51) | 17.21 (25.35)
  Change at Week 24: Bodily Pain | 11.68 (21.15) | 15.34 (24.39) | 14.23 (22.96) | 19.02 (24.36)
  Change at Week 24: Vitality | 3.21 (14.40) | 4.79 (15.75) | 3.17 (14.80) | 5.68 (14.56)
  Change at Week 24: Social Function | 4.95 (22.62) | 6.98 (25.53) | 7.69 (21.65) | 7.87 (18.02)
  Change at Week 24: Role Emotional | 4.44 (20.08) | 7.58 (23.56) | 6.41 (22.18) | 10.44 (25.25)
  Change at Week 24: Mental Health | 2.21 (12.30) | 1.23 (14.39) | 2.31 (13.24) | 2.11 (13.88)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Scores at Week 12, 24: Baseline Observation Carried Forward (BOCF)
Description: SF-36v2: standardized survey evaluating 8 domains of functional health and wellbeing (physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health). Total score for each domain were scaled 0 (poor health) to 100 (best health), higher scores indicating good health condition. For obtaining physical and mental component scores, z-score for each scale = (observed score - mean score for general 1990 United States [US] population)/corresponding standard deviation. The 2 component scores were obtained by multiplying each aspect z-score by physical or mental factor score coefficient (1990 general US population) and summing the eight products. Component scores indicated how many standard deviations higher (in case of positive z-score [better functioning])/lower (in case of negative z-score [worse functioning]) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
z-score
  Baseline: Mental Component Aggregate | 0.23 (1.08) | 0.21 (1.17) | 0.34 (1.11) | 0.30 (1.11)
  Baseline: Physical Component Aggregate | -1.79 (0.77) | -1.86 (0.73) | -1.89 (0.72) | -1.76 (0.76)
  Change at Week 12: Mental Component Aggregate | 0.16 (0.83) | 0.13 (0.98) | 0.14 (0.94) | 0.11 (0.90)
  Change at Week 12: Physical Component Aggregate | 0.37 (0.78) | 0.82 (0.95) | 0.80 (0.88) | 0.83 (0.85)
  Change at Week 24: Mental Component Aggregate | 0.07 (0.73) | 0.04 (0.94) | 0.06 (0.80) | 0.09 (0.83)
  Change at Week 24: Physical Component Aggregate | 0.38 (0.80) | 0.63 (0.89) | 0.55 (0.87) | 0.72 (0.90)

25. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 16
Population: Intent-to-treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo).
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 172 | 172 | 172 | 174
days | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events.

26. Secondary Outcome: Percentage of Participants Who Used Rescue Medications
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days per week could be taken as rescue medication.
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 154
percentage of participants
  Week 2 | 68.2 | 63.0 | 65.4 | 66.0
  Week 4 | 55.2 | 40.3 | 36.5 | 40.5
  Week 8 | 46.8 | 42.9 | 39.1 | 39.9
  Week 12 | 40.3 | 30.5 | 34.0 | 32.7
  Week 16 | 38.3 | 40.9 | 32.7 | 31.4
  Week 24 | 27.9 | 35.7 | 28.8 | 26.8

27. Secondary Outcome: Duration of Rescue Medication Use
Description: as for outcome 26
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 153
days
  Week 2 | 1.5 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 2.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0]
  Week 4 | 1.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 8 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 12 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 16 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 24 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]

28. Secondary Outcome: Amount of Rescue Medication Taken
Description: as for outcome 26
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 154 | 156 | 153
mg/week
  Week 2 | 3493.51 (4969.51) | 2818.18 (4063.15) | 3419.87 (4759.20) | 2993.46 (4226.71)
  Week 4 | 2691.56 (4484.61) | 1925.32 (3943.13) | 1891.03 (4038.24) | 2065.36 (4510.11)
  Week 8 | 2383.12 (4292.72) | 2133.12 (4199.69) | 1753.21 (4109.59) | 1934.64 (4568.45)
  Week 12 | 1941.56 (4184.45) | 1788.96 (4455.58) | 1567.31 (4359.67) | 1977.12 (6122.20)
  Week 16 | 2058.44 (4440.22) | 2207.79 (4696.58) | 1820.51 (4615.52) | 1663.40 (4367.50)
  Week 24 | 1704.55 (4183.54) | 1879.87 (4351.79) | 1836.54 (4768.57) | 1588.24 (4443.03)

ADVERSE EVENTS:
Description: Cases of osteonecrosis (ON) reported in this and other studies of this program, conducted up to 2010 were adjudicated post-hoc by an expert committee (2010-2012). Few of these events (2 of 87 reported ON cases), were confirmed as ON by the committee. Source: https://doi.org/10.1002/art.39492.
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Serious Adverse Events (participants affected / at risk) | 3/172 | 3/172 | 4/172 | 3/174
Other Adverse Events (participants affected / at risk) | 50/172 | 71/172 | 64/172 | 87/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=172) | Tanezumab 2.5 mg (N=172) | Tanezumab 5 mg (N=172) | Tanezumab 10 mg (N=174)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=172) | Tanezumab 2.5 mg (N=172) | Tanezumab 5 mg (N=172) | Tanezumab 10 mg (N=174)
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 2 | 4
Nausea (Gastrointestinal disorders) | 3 | 1 | 4 | 6
Fatigue (General disorders) | 0 | 4 | 4 | 3
Infusion related reaction (General disorders) | 1 | 0 | 1 | 4
Oedema peripheral (General disorders) | 1 | 3 | 6 | 11
Bronchitis (Infections and infestations) | 1 | 2 | 5 | 4
Nasopharyngitis (Infections and infestations) | 2 | 3 | 4 | 5
Sinusitis (Infections and infestations) | 0 | 4 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 10 | 11 | 7
Urinary tract infection (Infections and infestations) | 3 | 1 | 4 | 8
Contusion (Injury, poisoning and procedural complications) | 1 | 5 | 3 | 5
Fall (Injury, poisoning and procedural complications) | 3 | 6 | 5 | 7
Joint injury (Injury, poisoning and procedural complications) | 2 | 4 | 4 | 7
Blood creatine phosphokinase increased (Investigations) | 3 | 4 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 4 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 4
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 9
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 4
Carpal tunnel syndrome (Nervous system disorders) | 1 | 4 | 2 | 5
Dizziness (Nervous system disorders) | 3 | 3 | 4 | 7
Headache (Nervous system disorders) | 13 | 6 | 9 | 9
Hypoaesthesia (Nervous system disorders) | 2 | 7 | 5 | 6
Paraesthesia (Nervous system disorders) | 3 | 5 | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.